CLINICAL TRIAL: NCT06294782
Title: PrOsPective Cohort Study for STereotactic Arhythmia Radioablation (STAR) of Refractory Ventricular Tachycardia
Acronym: POPSTAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government); IRCCS Sacro Cuore Don Calabria di Negrar (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36/2022
Record Dates: First submitted 2022-05-10; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Refractory Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STereotactic Arhythmia Radioablation (STAR) (Experimental): Patients fulfilling the inclusion and exclusion criteria will undergo (or already underwent) a single-session 25 Gy STAR for the treatment of refractory monomorphic VT.
  Interventions: Radiation: STereotactic Arhythmia Radioablation (STAR)

INTERVENTIONS:
Radiation: STereotactic Arhythmia Radioablation (STAR) — STereotactic Arhythmia Radioablation (STAR)

SUMMARY:
This is a multicenter, interventional study. The study will enroll patients that fulfill the inclusion criteria over a 33-month period. Considering the small number of patients who will meet the study criteria, it is also possible to include retrospective patients who already underwent STAR (for instance, as part of a compassionate program) if they meet all the inclusion and exclusion criteria as well as the treatment planning standardized requirements and sign their consent to this trial. All patients prospectively enrolled will undergo a flow of investigations following a standardized approach. ICD programming will be standardized.

ELIGIBILITY:
Inclusion Criteria:

1. Structural heart disease (SHD) defined as left ventricular dysfunction (LVEF < 55%), or right ventricular dysfunction (FAC <35%) or presence of ventricular scar, pathological hypertrophy, wall bulging or inflammatory conditions.
2. Optimized medical treatment for the underlying SHD
3. ICD or CRT-D recipient
4. ≥ 1 episodes of sustained or treated (with either anti-tachycardia pacing or shock, internal or external) monomorphic VT (MMVT) resistant to at least one invasive VT ablation attempt, unless contraindicated or deemed at high risk. Reason for lack of ablation must be specified

Exclusion Criteria:

1. Age < 18 or > 85 years.
2. Inability to provide informed consent.
3. Acute myocardial infarction or recent primary coronary intervention or cardiac surgery (<3 months)
4. Primary electrical disease (e.g. long QT syndrome, short QT syndrome, catecholaminergic polymorphic ventricular tachycardia, Brugada syndrome).
5. Reversible and/or treatable cause of VT (e.g., drug-induced or intoxication)
6. ICD electrode malfunction or ICD readings outside reference range
7. Pregnancy or breast feeding
8. Patients with polymorphic VT/VF

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
VT storm and incessant VT | 6 months
  6-month survival free from VT storm (3 or more episodes or sustained or treated VT within 24 hours) and incessant VT (binary endpoint), including an initial blanking period of 8 weeks.
adverse events | 33 months
  : measured by registered adverse events using the CTCAE v5 system, 'early' (up to 30 days), 'intermediate' (30-90 days), and 'late' (>90 days after treatment). The extensive mandatory and optional follow-up examinations provide the basis for detecting these adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Turin, Turin, Italy